CLINICAL TRIAL: NCT02284425
Title: Study of REGN1193 in Patients With Type 2 Diabetes Mellitus
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R1193-DM-1402
Record Dates: First submitted 2014-10-22; First posted 2014-11-06 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — crotedumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part A (Experimental): Participants in Part A will consist of 4 sequential ascending dose cohorts. Each cohort will receive 1 of 4 ascending dose levels of study drug (REGN1193) or placebo.
  Interventions: Drug: REGN1193; Drug: Placebo
- Part B (Experimental): Participants in Part B will consist of a single cohort and will receive three doses of study drug (REGN1193) or placebo.
  Interventions: Drug: REGN1193; Drug: Placebo

INTERVENTIONS:
Drug: REGN1193
Drug: Placebo

SUMMARY:
This is a phase 1, randomized, double-blind, placebo-controlled study to evaluate the safety and tolerability of REGN1193 in patients with Type 2 Diabetes Mellitus.

ELIGIBILITY:
Inclusion Criteria:

1. Metformin monotherapy at a dose of ≥1000 mg/day (up to the maximum daily dose of 2550 mg per day) for ≥8 weeks prior to randomization
2. Hemoglobin A1c value of ≥7.0% to ≤10.0%
3. Fasting plasma glucose value ≥130 mg/dL and ≤240 mg/dL

Exclusion Criteria:

1. Type 1 diabetes mellitus
2. Use of insulin or oral or injectable antihyperglycemic medications during the 8 weeks prior to randomization
3. A severe hypoglycemic event in the 6 months prior to randomization

Note: The eligibility criteria listed above is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial therefore not all inclusion/ exclusion criteria are listed.

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2014-10; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of treatment emergent adverse events (TEAEs) | Day 1 through Day 57

SECONDARY OUTCOMES:
Pharmacodynamic profile of REGN1193 as measured by plasma glucose over time | Day 1 through Day 57
Concentration of REGN1193 in serum over time | Day 1 through Day 57

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (3):
- United States (3):
  - Miami, Florida
  - Atlanta, Georgia
  - Knoxville, Tennessee